CLINICAL TRIAL: NCT02122588
Title: OVArian Cancer Non-Interventional Study. Treatment hAbits and Epidemiology of BRCA in Russian Federation - OVATAR
Brief Title: OVArian Cancer Non-Interventional Study - OVATAR
Acronym: OVATAR
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: RUSSCO (Russian Society of Clinical Oncology) (Unknown)
Responsible Party: Sponsor
Other Study IDs: NIS-ORU-XXX-2014/1
Record Dates: First submitted 2014-04-23; First posted 2014-04-24 (Estimated); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Ovarian, Peritoneal, Fallopian Tube Cancer, BRCAm+ in Russia
Keywords: serous and endometrioid ovarian, peritoneal, fallopian tube cancer, hereditary ovarian cancer, BRCA (breast cancer gene) mutation, genetic testing
MeSH Terms: conditions — Fallopian Tube Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- OVATAR study patients: Females with serous and endometrioid ovarian, peritoneal and fallopian tube cancer 18 years and older, diagnosed 3 months before enrolment into the study or later, consented to participate in this non-interventional study, who are being treated for OC, FTC (Fallopian Tube Cancer) and PC (Peritoneal Cancer) in the oncology hospitals/departments in the Russian Federation.

SUMMARY:
This is a multicentre, non-interventional, prospective study to be carried out in representative hospitals in order to assess 1st line treatment management and diagnostic approaches applied to ovarian, peritoneal and fallopian tube cancer management in Russia and assess patients' characteristics and the occurrence of BRCA (Breast Cancer gene) mutations among Russian women with serous and endometrioid ovarian, peritoneal and fallopian tube cancer. No additional procedures besides those already used in the routine clinical practice will be applied to the patients. Treatment assignment will be done according to the current practice.

DETAILED DESCRIPTION:
This is a multicentre, non-interventional, prospective study to be carried out in representative hospitals in order to assess ovarian, fallopian tube and peritoneal cancer management in Russia. No additional procedures besides those already used in the routine clinical practice will be applied to the patients. Treatment assignment will be done according to the current practice.

It is planned to enrol 300 subjects in up to 30 sites in Russian Federation. The average number of patients per site is planned as 10-15; there are no restrictions on minimum and maximum number of subjects per site in this study.

The disease treatments approaches in 1st line treatment of serous and endometrioid ovarian, peritoneal and fallopian tube cancer (both chemotherapy and surgery) is considered as the primary outcome variable in this study.

Along with other diagnosis examinations the analysis of frequent mutations in the gen BRCA1 (5382insC, 4154delA, 185delAG and C61G (c.300T>G)) will be performed by local or regional laboratories.

Those patients with BRCAm+ OC (Ovarian Cancer) will be observed prospectively during 2 years after the baseline visit or till progression at the 1st line treatment with regards to OC treatment details and outcomes. The patients for whom BRCA mutations not found will participate in the baseline assessments only and will not be followed up. Accordingly, 1 study visit (screening/baseline) is planned for all patients and 1 FU visit (Year 2) is planned for BRCAm+ patients.

The subpopulation of the patients with the congenital serous and endometrioid ovarian, peritoneal and fallopian tube cancer with the corresponding family history will undergo the broadened genetic testing panel (sequencing of all coding areas of genes BRCA1 and BRCA2).

Information regarding patient demographics, the disease characteristics, management approaches, diagnostic tests performed and medication received by the patient will be taken from the medical records.

ELIGIBILITY:
Inclusion Criteria:

1. The voluntary obtained informed consent signed by both the subject and the investigator.
2. Confirmed serous and endometrioid ovarian cancer or fallopian tube cancer or peritoneal cancer diagnosed 3 months before enrolment into the study or later
3. Patients on treatment for OC (Ovarian Cancer) or FTC (Fallopian Tube Cancer) or PC (Peritoneal Cancer)

Exclusion Criteria:

1. The ovarian cancer histology other than serous and endometrioid.
2. Patients participating in clinical studies.
3. Any medical condition which on the opinion of the investigator may interfere the patient's participation in the trial.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Females with serous and endometrioid ovarian, peritoneal and fallopian tube cancer 18 years and older, diagnosed 3 months before enrolment into the study or later, consented to participate in this non-interventional study, who are being treated for OC, FTC and PC in the oncology hospitals/departments in the Russian Federation.
Sampling Method: Non-Probability Sample
Enrollment: 503 (Actual)
Dates: Start 2014-06-30 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of 1st line chemotherapy treatment of serous and endometrioid ovarian, peritoneal and fallopian tube cancer (drugs by INN (International Nonproprietary Name), doses, regimen) | up to 14 months
  Evaluation of 1st line chemotherapy treatment of serous and endometrioid ovarian, peritoneal and fallopian tube cancer (drugs by INN, doses, regimen)

SECONDARY OUTCOMES:
Data collection of patients characteristics (gender, age, race, co-morbidities, family history of ovarian and breast cancer) | up to 14 months
  Data collection of patients characteristics (gender, age, race, co-morbidities, family history of ovarian and breast cancer)
Data collection of disease information (including genetic testing results) | up to 14 months
  Data collection of disease information (including genetic testing results)
Proportion of BRCAm+ among serous and endometrioid ovarian, peritoneal and fallopian tube cancer in Russia. | up to 14 months
  Proportion of BRCAm+ among serous and endometrioid ovarian, peritoneal and fallopian tube cancer in Russia.
Evaluation of response to 1st line chemotherapy treatment of serous and endometrioid BRCAm+ ovarian, peritoneal and fallopian tube cancer | up to 3 months
  Evaluation of response to 1st line chemotherapy treatment of serous and endometrioid BRCAm+ ovarian, peritoneal and fallopian tube cancer
Assessment of relapses after 1st line of Pt (Platinum)-containing regimen for BRCAm+ patients | up to 3 months
  Assessment of relapses after 1st line of Pt-containing regimen for BRCAm+ patients
Evaluation of 2nd line chemotherapy treatment of serous and endometrioid ovarian, peritoneal and fallopian tube cancer (drugs by INN, doses, regimen) for BRCAm+ patients who have progressed after 1st line chemotherapy | up to 3 months
  Evaluation of 2nd line chemotherapy treatment of serous and endometrioid ovarian, peritoneal and fallopian tube cancer (drugs by INN, doses, regimen) for BRCAm+ patients who have progressed after 1st line chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Karin Otter, Study Director — AstraZeneca; Vera Gorbunova, Principal Investigator — Russian Cancer Research Center named after NN Blokhin; Alexandra Tyulandina, Principal Investigator — Russian Cancer Research Center named after NN Blokhin; Larisa Kolomietz, Study Chair — Research Oncology Center, Tomsk; Tatiana Kekeeva, Study Chair — Research Centre for Medical Genetics, Moscow
Locations (22):
- Russia (22):
  - Research Site, Arkhangelsk
  - Research Site, Chelyabinsk
  - Research Site, Irkutsk
  - Research Site, Izhevsk
  - Research Site, Kaluga
  - Research Site, Khabarovsk
  - Research Site, Moscow
  - Research Site, Novorossiysk
  - Research Site, Novosibirsk
  - Research Site, Obninsk
  - Research Site, Omsk
  - Research Site, Orenburg
  - Research Site, Pyatigorsk
  - Research Site, Rostov-on-Don
  - Research Site, Saint Petersburg
  - Research Site, Samara
  - Research Site, Sochi
  - Research Site, Tomsk
  - Research Site, Tula
  - Research Site, Tver'
  - Research Site, Ufa
  - Research Site, Vladimir

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=2948&filename=Ovatar_Observational%20Study%20Report_synopsis.pdf